CLINICAL TRIAL: NCT02037893
Title: A Four-arm, Randomized, Double-blind, Active and Placebo Controlled Study to Determine the Safety and Efficacy of a Combination Antipyrine and Benzocaine Otic Solution Compared With Antipyrine Otic Solution Alone, Benzocaine Otic Solution Alone and to Placebo Otic Solution to Relieve Pain Symptoms in Children With Acute Otitis Media.
Brief Title: Four Arm Safety & Efficacy With Antipyrine and Benzocaine Otic Solution in Children With Acute Otitis Media
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Currax Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: PNX-CL-001
Record Dates: First submitted 2014-01-13; First posted 2014-01-16 (Estimated); Results first posted 2018-08-31 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2018-08

CONDITIONS: Acute Otitis Media
MeSH Terms: conditions — Otitis Media | interventions — Antipyrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Antipyrine and Benzocaine Otic solution (Experimental): antipyrine 54 mg and benzocaine 14 mg. Apply drops along the wall of the ear canal until filled and repeating every 3 hours for 24 hours unless the subject is sleeping
  Interventions: Drug: Antipyrine and Benzocaine otic solution; Drug: Placebo Otic solution
- Antipyrine Otic Solution (Active Comparator): Antipyrine 54 mg and glycerine dehydrated to 1.0 mL. Apply drops along the wall of the ear canal until filled and repeating every 3 hours for 24 hours unless the subject is sleeping
  Interventions: Drug: Antipyrine Otic Solution; Drug: Placebo Otic solution
- Benzocaine Otic Solution (Active Comparator): benzocaine 14 mg and glycerine dehydrated to 1.0 ml. Apply drops along the wall of the ear canal until filled and repeating every 3 hours for 24 hours unless the subject is sleeping
  Interventions: Drug: Benzocaine Otic Solution; Drug: Placebo Otic solution
- Placebo (Placebo Comparator): Placebo otic solution will be glycerin that is dehydrated . Apply drops along the wall of the ear canal until filled and repeating every 3 hours for 24 hours unless the subject is sleeping
  Interventions: Drug: Placebo Otic solution

INTERVENTIONS:
Drug: Antipyrine and Benzocaine otic solution — antipyrine 54 mg and benzocaine 14 mg
  Arms: Antipyrine and Benzocaine Otic solution
Drug: Antipyrine Otic Solution — Antipyrine 54 mg and glycerine dehydrated to 1.0 mL
  Arms: Antipyrine Otic Solution
Drug: Benzocaine Otic Solution — benzocaine 14 mg and glycerine dehydrated to 1.0 mL
  Arms: Benzocaine Otic Solution
Drug: Placebo Otic solution — Placebo otic solution will be glycerin that is dehydrated

SUMMARY:
The primary objective is to compare the effect of treatment with a combination of ear solutions on the reduction of pain symptoms at 1 hour after dosing in children with acute otitis media.

DETAILED DESCRIPTION:
Reduction of pain symptoms will be measured by using the Face, Legs, Activity, Cry, Consolability Scale (FLACC) and the Faces pain Scale Revised (FPS-R).

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of Acute Otitis Media
* Moderate to severe pain
* Normally active and in good health as determined by the PI
* Parent or legal guardian consent
* Caregiver available to complete diaries during study

Exclusion Criteria:

* History of or current Perforated tympanic membrane
* Tympanostomy tubes
* Acute or chronic otitis externa
* seborrheic dermatitis
* Received any otic topical or systemic antibiotic within 14 days of enrollment
* Receiving medication on a chronic basis for pain
* Known hypersensitivity to investigational product.
* clinical significant mental illness as determined by the PI
* Exposed to another investigational agent within 30 days before study entry. Any condition the PI believed will interfere with the ability to comply with all study procedures
* History of glucose 6-phosphate dehydrogenase deficiency
* History or currently anemic
* Congenital methemoglobinemia
* Recent history of acute gastroenteritis within 14 days of enrollment

Ages: 2 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 112 (Actual)
Dates: Start 2013-11; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Goldberg, MD, Principal Investigator — Visions Clinical Research; Gerald Shockey, MD, Principal Investigator — Desert Clinical Research; Shane Christensen, MD, Principal Investigator — Foothill Family Clinic South; Stephanie Plunkett, MD, Principal Investigator — First Med East; Katie Julien, MD, Principal Investigator — Jordan River Family Medcine; James Peterson, MD, Principal Investigator — Foothill Family Clinic; John Ansely, MD, Principal Investigator — Carolina Ear, Nose and Throat Clinic; James Hendrick, MD, Principal Investigator — Kentucky Pediatric and Adult Research; Amy Agua, MD, Principal Investigator — Visions Clinical Research Boyton Beach; Bryan Harvey, MD, Principal Investigator — Childrens Investigational Research Program
Locations (10):
- United States (10):
  - Desert Clinical Research, Mesa, Arizona
  - Visions Clinical Research, Tucson, Arizona
  - Childrens Investigational Research Program, Bentonville, Arkansas
  - Visions Clinical Research, Boynton Beach, Florida
  - Kentucky Pediatric and Adult Research, Bardstown, Kentucky
  - Carolina Ear, Nose and Throat Clinic, Orangeburg, South Carolina
  - Foothill Family Clinic, Salt Lake City, Utah
  - FirstMed East, Salt Lake City, Utah
  - Foothill Family Clinic South, Salt Lake City, Utah
  - Jordan River Family Medicine, South Jordan, Utah

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Antipyrine and Benzocaine Otic Solution | Antipyrine Otic Solution | Benzocaine Otic Solution | Placebo
Started | 32 | 25 | 27 | 28
Completed | 32 | 25 | 26 | 28
Not Completed | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Antipyrine and Benzocaine Otic Solution | Antipyrine Otic Solution | Benzocaine Otic Solution | Placebo | Total
Number analyzed (Participants) | 32 | 25 | 27 | 28 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.4 (3.27) | 4.4 (3.36) | 4.5 (3.75) | 3.5 (3.35) | 4.2 (3.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 11 | 10 | 44
  Male | 19 | 15 | 16 | 18 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 6 | 5 | 6 | 26
  Not Hispanic or Latino | 23 | 19 | 21 | 22 | 85
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Black or African American | 5 | 2 | 2 | 3 | 12
  White | 24 | 22 | 24 | 24 | 94
  More than one race | 2 | 1 | 1 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 32 | 25 | 27 | 28 | 112

OUTCOME MEASURES:

1. Primary Outcome: Face, Legs, Activity, Cry, Consolability Scale (FLACC) or Faces Pain Scale Revised (FPS-R)
Description: The FLACC was completed by the caregiver to assess pain intensity for subjects aged 2 months to less than 5 years. The FLACC consists of five domains that are rated as 0, 1, or 2 (total scores range from 0 to 10). A lower score indicates lower level of pain.
  The FPS-R was completed by the subject aged 5 to 12 years. For this assessment, the subject selected the pain intensity by using faces that show increasing discomfort. Total scores range from 0 to 10. A lower score indicates lower level of pain.
Time Frame: Baseline and 1 hour after a single dose
Population: Intent-to-Treat population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Antipyrine and Benzocaine Otic Solution | Antipyrine Otic Solution | Benzocaine Otic Solution | Placebo
Number analyzed (Participants) | 30 | 24 | 22 | 27
units on a scale | -4.3 (3.43) | -5.0 (2.82) | -4.6 (2.97) | -4.9 (2.13)

2. Secondary Outcome: Face, Legs, Activity, Cry, Consolability Scale (FLACC) or Faces Pain Scale Revised (FPS-R)15 Min Post First Dose
Description: The relative change from baseline in pain intensity as measured by changes in FLACC scores or FPS-R scores between baseline and 15 and 30 minutes, and 3, 6, 12, 24, 36, 48, 60, and 72 hours after first dose.
  The FLACC was completed by the caregiver to assess pain intensity for subjects aged 2 months to less than 5 years. The FLACC consists of five domains that are rated as 0, 1, or 2 (total scores range from 0 to 10). A lower score indicates lower level of pain.
  The FPS-R was completed by the subject aged 5 to 12 years. For this assessment, the subject selected the pain intensity by using faces that show increasing discomfort. Total scores range from 0 to 10. A lower score indicates lower level of pain.
Time Frame: Change from Baseline to 15 min post first dose
Population: The intent-to-treat (ITT) population included all subjects who were randomized to receive treatment and had at least one postscreening efficacy assessment at the timepoint of interest.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Antipyrine and Benzocaine Otic Solution | Antipyrine Otic Solution | Benzocaine Otic Solution | Placebo
Number analyzed (Participants) | 31 | 24 | 24 | 28
units on a scale | -3.6 (0.48) | -3.6 (0.54) | -3.4 (0.51) | -3.8 (0.51)

3. Secondary Outcome: Face, Legs, Activity, Cry, Consolability Scale (FLACC) or Faces Pain Scale Revised (FPS-R) 30 Min Post First Dose
Description: as for outcome 2
Time Frame: Change from Baseline to 30 min post first dose
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Antipyrine and Benzocaine Otic Solution | Antipyrine Otic Solution | Benzocaine Otic Solution | Placebo
Number analyzed (Participants) | 30 | 24 | 24 | 27
units on a scale | -3.9 (0.45) | -4.3 (0.51) | -4.4 (0.49) | -4.8 (0.48)

4. Secondary Outcome: Face, Legs, Activity, Cry, Consolability Scale (FLACC) or Faces Pain Scale Revised (FPS-R) 3 Hour Post First Dose
Description: as for outcome 2
Time Frame: Change from Baseline to 3 hour post first dose
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Antipyrine and Benzocaine Otic Solution | Antipyrine Otic Solution | Benzocaine Otic Solution | Placebo
Number analyzed (Participants) | 29 | 22 | 20 | 23
units on a scale | -3.4 (0.47) | -3.9 (0.53) | -3.8 (0.50) | -3.5 (0.50)

5. Secondary Outcome: Face, Legs, Activity, Cry, Consolability Scale (FLACC) or Faces Pain Scale Revised (FPS-R) 6 Hours Post First Dose
Description: as for outcome 2
Time Frame: Change from Baseline to 6 hour post first dose
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Antipyrine and Benzocaine Otic Solution | Antipyrine Otic Solution | Benzocaine Otic Solution | Placebo
Number analyzed (Participants) | 27 | 21 | 19 | 19
units on a scale | -3.4 (0.50) | -4.0 (0.56) | -3.9 (0.54) | -3.8 (0.54)

6. Secondary Outcome: Face, Legs, Activity, Cry, Consolability Scale (FLACC) or Faces Pain Scale Revised (FPS-R) 12 Hours Post First Dose
Description: as for outcome 2
Time Frame: Change from Baseline to 12 hour post first dose
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Antipyrine and Benzocaine Otic Solution | Antipyrine Otic Solution | Benzocaine Otic Solution | Placebo
Number analyzed (Participants) | 19 | 16 | 17 | 14
units on a scale | -3.9 (0.53) | -4.3 (0.60) | -4.1 (0.57) | -4.0 (0.57)

7. Secondary Outcome: Face, Legs, Activity, Cry, Consolability Scale (FLACC) or Faces Pain Scale Revised (FPS-R) 24 Hours Post First Dose
Description: as for outcome 2
Time Frame: Change from Baseline to 24 hour post first dose
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Antipyrine and Benzocaine Otic Solution | Antipyrine Otic Solution | Benzocaine Otic Solution | Placebo
Number analyzed (Participants) | 29 | 20 | 21 | 22
units on a scale | -5.5 (0.42) | -4.4 (0.48) | -4.2 (0.46) | -4.6 (0.46)

8. Secondary Outcome: Face, Legs, Activity, Cry, Consolability Scale (FLACC) or Faces Pain Scale Revised (FPS-R) 36 Hours Post First Dose
Description: as for outcome 2
Time Frame: Change from Baseline to 36 hour post first dose
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Antipyrine and Benzocaine Otic Solution | Antipyrine Otic Solution | Benzocaine Otic Solution | Placebo
Number analyzed (Participants) | 22 | 20 | 19 | 20
units on a scale | -5.5 (0.42) | -4.6 (0.48) | -4.4 (0.46) | -5.5 (0.45)

9. Secondary Outcome: Face, Legs, Activity, Cry, Consolability Scale (FLACC) or Faces Pain Scale Revised (FPS-R) 48 Hours Post First Dose
Description: as for outcome 2
Time Frame: Change from Baseline to 48 hour post first dose
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Antipyrine and Benzocaine Otic Solution | Antipyrine Otic Solution | Benzocaine Otic Solution | Placebo
Number analyzed (Participants) | 30 | 23 | 22 | 26
units on a scale | -5.4 (0.37) | -5.3 (0.42) | -4.7 (0.40) | -5.9 (0.40)

10. Secondary Outcome: Face, Legs, Activity, Cry, Consolability Scale (FLACC) or Faces Pain Scale Revised (FPS-R) 60 Hours Post First Dose
Description: as for outcome 2
Time Frame: Change from Baseline to 60 hour post first dose
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Antipyrine and Benzocaine Otic Solution | Antipyrine Otic Solution | Benzocaine Otic Solution | Placebo
Number analyzed (Participants) | 24 | 21 | 19 | 20
units on a scale | -5.4 (0.33) | -5.4 (0.37) | -5.4 (0.36) | -6.2 (0.36)

11. Secondary Outcome: Face, Legs, Activity, Cry, Consolability Scale (FLACC) or Faces Pain Scale Revised (FPS-R) 72 Hours Post First Dose
Description: as for outcome 2
Time Frame: Change from Baseline to 72 hour post first dose
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Antipyrine and Benzocaine Otic Solution | Antipyrine Otic Solution | Benzocaine Otic Solution | Placebo
Number analyzed (Participants) | 30 | 24 | 24 | 26
units on a scale | -5.9 (0.29) | -5.9 (0.33) | -5.4 (0.32) | -6.1 (0.32)

ADVERSE EVENTS:
Time Frame: Up to 120 hours after first dose
Arm/Group | Antipyrine and Benzocaine Otic Solution | Antipyrine Otic Solution | Benzocaine Otic Solution | Placebo
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/25 | 0/27 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/25 | 0/27 | 0/28
Other Adverse Events (participants affected / at risk) | 6/32 | 9/25 | 4/27 | 5/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antipyrine and Benzocaine Otic Solution (N=32) | Antipyrine Otic Solution (N=25) | Benzocaine Otic Solution (N=27) | Placebo (N=28)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoacisis (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (4) | 1 (1) | 0 (0)
Application site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lice infestation (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis Media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Otitis Media acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral rash (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No